CLINICAL TRIAL: NCT04897893
Title: Impact of a Daily Supplementation With 2.0g of Eicosapentaenoic Acid Monoglycerids (MAG-EPA) on the Arachidonic and Eicosapentaenoic Acids Ratio (AA/EPA) and on Blood Inflammation Markers in a Healthy Population Aged of 50 and Older.
Brief Title: Impact of 2.0g Daily of MAG-EPA on the AA/EPA Ratio and Inflammation Biomarkers in a Healthy Population Aged of 50+.
Acronym: IO3-04
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SCF Pharma (Industry)
Collaborators: Integrated Health and Social Services Centres (CISSS) de la Gaspésie (Unknown); Integrated Health and Social Services Centres (CISSS) du Bas-St-Laurent (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IO3-04
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Inflammation
Keywords: COX-2, Inflammation, MAG-EPA
MeSH Terms: conditions — Inflammation | interventions — 1-eicosapentaenoylglycerol

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, phase IV pilot study where all participants receive the same treatment for a similar duration. Their pre-treatment baseline condition will serve as a comparator for the effects observed following MAG-EPA treatment. There is no control group in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): All subjects enrolled in the study will receive an identical dose of 2g/day (4 capsules of MAG-EPA) which will be taken by the subject at home. The duration of treatment should not be prolonged in the event of missed doses, that is, treatment should end on the 84th day as planned. A deviation of ± 3 days is acceptable, which means that treatment can be stopped from day 81 to day 87 of subject's participation.
  Interventions: Other: Eicosapentaenoic acid monoglycerid (MAG-EPA)

INTERVENTIONS:
Other: Eicosapentaenoic acid monoglycerid (MAG-EPA) — MAG-EPA is an omega-3 fatty acid classified in canada as a Natural Health Product (NHP). The NHP is approuved under the Natural Health Product number (NPN # 80050187).

SUMMARY:
According to scientific literature, oils containing omega-3 fatty acids may decrease certain risk factors for cardiovascular disease such as blood pressure, blood level of triglycerides (TGs) and cholesterol. The omega-3 index (amount of EPA + DHA in the blood) is a recognized biomarker for assessing risk factors for cardiovascular disease. Its optimal value is 8% compared to the Canadian population average of only 4.5%. The scientific literature contains several good studies on omega-3 fatty acids, however, it is difficult to compare dose-response relationships between studies since formulations are not similar and markers of exposure to treatment are not standardized. The AA/EPA ratio, combined with the omega-3 index, is a good way to monitor the increase in omega-3 levels in the blood, but especially to determine the inflammatory status of a patient. Indeed, eicosapentaenoic acid (EPA) is a fatty acid with inflammation-resolving properties, while arachidonic acid (AA) is a pro-inflammatory agent. A high AA/EPA ratio therefore indicates a high inflammatory status while a low ratio indicates a better balance between active inflammation and its resolution. Moreover, it was published in 2018 that a AA/EPA ratio of around 3 was directly associated with a 25% reduction in the relative risk of cardiovascular disease. Therefore, the investigator wants to determine the minimum MAG-EPA dose needed to achieve an AA/EPA ratio equivalent to 4g of EPA in the form of ethyl ester (EE-EPA). It is reasonable to estimate that 2g of MAG-EPA should be sufficient to produce an average AA/EPA ratio around 3.1.

DETAILED DESCRIPTION:
This pilot study aims to determine the average value of the ratio of arachidonic to eicosapentaenoic acids (AA/EPA) in a population aged 50 and over without any particular medical condition when supplemented with 2g per day of MAG-EPA for 12 weeks.

1.1 Main objectives

1. To recruit a population of 30 subjects aged 50 and over without any particular medical condition in order to administer 2.0g of MAG-EPA per day for 12 weeks.
2. By measuring the omega-3 index level of all subjects before starting the study and thereafter every 6 weeks over a total period of 12 weeks, the investigator will analyse the individual levels of arachidonic acids and eicosapentaenoic acids to establish the AA/EPA ratio at each visit.
3. The initial AA/EPA ratio will be compared to that obtained after 12 weeks of MAG-EPA supplementation. The results of the present study will be compared to those obtained by daily supplementation with 4.0g of EE-EPA over a similar period of time (taken from the scientific literature) to determine whether MAG-EPA meets the statistical criteria for non- inferiority in terms of response to the AA/EPA ratio.

1.2 Secondary objectives

1. Analyze markers of inflammation such as CRP and PSA (in men only) as well as COX-2 activity before starting the study and thereafter every 6 weeks for a total period of 12 weeks in order to identify the best clinical markers of response to MAG-EPA in the context of the treatment of inflammation.
2. Analyze the lipid profile, before starting the study and thereafter every 6 weeks over a total period of 12 weeks in order to better characterize the effects of MAG-EPA supplementation on this clinical parameter.
3. Determine the proportion of participants who achieve an omega-3 index of at least 8%.
4. Characterize the effects of MAG-EPA supplementation on the proportion of senescent white blood cells, on the omega-6/omega-3 ratio as well as on the subject's blood trans fat content.

ELIGIBILITY:
Inclusion Criteria:

1. Participant aged 50 or over.
2. Available for the entire duration of the study and willing to participate based on the information provided in the ICF duly read and signed by the latter.
3. Participant not presenting any intellectual problems likely to limit the validity of the consent to participate in the study and the respect of protocol requirements, having the capacity to cooperate adequately, to understand and to follow the instructions of the doctor or his delegates.
4. Participant who has no difficulty swallowing tablets or capsules.

Exclusion Criteria:

1. Known allergy or intolerance to fish or history of allergic reactions attributable to fish, or to a compound similar to fish oil.
2. Pregnant or breastfeeding woman.
3. Participant who used omega-3 supplements within 60 days of study day 1.
4. Difficulty obtaining blood samples by capillary or venous puncture at the time of selection.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Fatty acids profile analysis | 12 weeks
  The individual content of all fatty acids present in humans will be analysed for each subject on red blood cells obtained by blood sampling after 6 and 12 weeks of supplementation with eicosapentaenoic acid monoglycerides (MAG-EPA). With the individual fatty acid contents obtained for each timepoint, it will be possible to calculate an omega-3 index (% of omega-3, EPA + DHA, on total fatty acids), the total omega-6/omega-3 ratio and finally, the ratio of arachidonic acids to eicosapentaenoic acids (AA/EPA).

SECONDARY OUTCOMES:
Research of clinical biomarkers for inflammation. | 12 weeks
  For each timepoint (0, 6 and 12 weeks), PSA (for men only) and CRP will be analysed through the health services laboratories. The activity of the COX-2 protein will also be analysed in Dr Fortin's research laboratory. The results at 6 and 12 weeks will be compared to the baseline analysis to evaluate the potential in resolution of inflammation when subjects are supplemented with 2.0g daily of MAG-EPA.
Proportion of subjects with a 8% or higher omega-3 index after 12 weeks of supplementation | 12 weeks
  The omega-3 index will be analysed for all subjects included in the study after 6 and 12 weeks of supplementation with 2.0g of MAG-EPA. The proportion of subjects with an omega-3 index equal or higher to 8% will be calculated at this dose for the 12 weeks timepoint.
Impact of supplementation on proportion of senescent white blood cells. | 12 weeks
  At each study visit (week 0, 6 and 12), a whole blood sample will be sent to the laboratory of Dr Fortin for a flow cytometry analysis. The proportion of senescent white blood cells at last visit will be compared to the proportion obtained at baseline.
Comparison of pre and post-dose Lipid profile. | 12 weeks
  At each study visit (week 0, 6 and 12), a whole blood sample will be sent to the health services laboratory for a lipid profile analysis. The results at last visit will be compared to those obtained at baseline and week 6 to detect any change caused by supplementation.
Obsevation and research of any adverse events | 16 weeks
  Subjects will be questionned about any changes in their health status at each study visit (week 0, week 6 and week 12). A telephone follow-up will be done halfway between visits (week 3 and week 9).They will also be instructed to note and report any change in their health status between follow-ups. For each adverse event, the following will be noted: start date, time and severity; end date, time, maximal severity and outcome; seriousness, causal relationship to study drug and expectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C Fortin, PhD, Principal Investigator — SCF Pharma
Locations (2):
- Canada (2):
  - SCF Pharma, Maria, Quebec
  - SCF Pharma, Rimouski, Quebec